CLINICAL TRIAL: NCT02956044
Title: A Phase 1, Open-label, Randomized, Three-period, Crossover Study to Evaluate Pharmacokinetic Interaction Between Bexagliflozin Tablets and Metformin, Glimepiride, or Sitagliptin in Healthy Subjects
Brief Title: Interaction of Bexagliflozin With Metformin, Glimepiride and Sitagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-453
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — bexagliflozin; Metformin; glimepiride; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Group 1: Bexagliflozin alone (Active Comparator)
  Interventions: Drug: Bexagliflozin
- Group 1: Metformin alone (Active Comparator)
  Interventions: Drug: Metformin
- Group 1: Bexagliflozin + Metformin (Active Comparator)
  Interventions: Drug: Bexagliflozin; Drug: Metformin
- Group 2: Bexagliflozin alone (Active Comparator)
  Interventions: Drug: Bexagliflozin
- Group 2: Glimepiride alone (Active Comparator)
  Interventions: Drug: Glimepiride
- Group 2: Bexagliflozin + Glimepiride (Active Comparator)
  Interventions: Drug: Bexagliflozin; Drug: Glimepiride
- Group 3: Bexagliflozin alone (Active Comparator)
  Interventions: Drug: Bexagliflozin
- Group 3: Sitagliptin alone (Active Comparator)
  Interventions: Drug: Sitagliptin
- Group 3: Bexagliflozin + Sitagliptin (Active Comparator)
  Interventions: Drug: Bexagliflozin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablets, 20 mg
  Arms: Group 1: Bexagliflozin + Metformin; Group 1: Bexagliflozin alone; Group 2: Bexagliflozin + Glimepiride; Group 2: Bexagliflozin alone; Group 3: Bexagliflozin + Sitagliptin; Group 3: Bexagliflozin alone
Drug: Metformin — 1000 mg metformin
  Arms: Group 1: Bexagliflozin + Metformin; Group 1: Metformin alone
Drug: Glimepiride — 4 mg glimepiride
  Arms: Group 2: Bexagliflozin + Glimepiride; Group 2: Glimepiride alone
Drug: Sitagliptin — 100 mg sitagliptin
  Arms: Group 3: Bexagliflozin + Sitagliptin; Group 3: Sitagliptin alone

SUMMARY:
The purpose of this study is to examine the drug-drug interaction in your body when given the study drug, bexagliflozin, with three commonly used ant-diabetic medications, metformin, glimepiride or sitagliptin. The study will also evaluate how safe the study drug is and how well the study drug is tolerated when taken with metformin, glimepiride or sitagliptin.

DETAILED DESCRIPTION:
A total of 54 healthy subjects were enrolled and assigned to one of three groups of eighteen. Each group participated in one of three open-label, randomized, three treatment period, crossover studies:

* Group 1: Bexagliflozin/metformin drug-drug interaction (DDI)
* Group 2: Bexagliflozin/glimepiride DDI
* Group 3: Bexagliflozin/sitagliptin DDI For each Group, every subject received a single dose of bexagliflozin tablet, 20 mg, alone, a single dose of an oral hypoglycemic agent (OHA) (1000 mg metformin, 2 mg glimepiride, or 100 mg sitagliptin) alone, and the combination of both (bexagliflozin tablet and OHA) alternately in a crossover fashion, with three treatment periods separated by a washout period of at least 7 days. Within each Group, subjects were randomized to one of six treatment sequences in an equal ratio.

To prevent hypoglycemia, subjects assigned to Group 2 (bexagliflozin/glimepiride DDI) received approximately 300 mL of a solution containing 50 g of glucose with study medication at the time of dosing, as well as approximately 75 mL of a solution containing 12.5 g of glucose every 15 minutes for 4 hours post-dose.

For each treatment period in Group 1 (bexagliflozin/metformin DDI) and Group 2 (bexagliflozin/glimepiride DDI), subjects were admitted to the clinic on the day before dosing and stayed in the clinic until 48 h post-dose. For Group 3 (bexagliflozin/sitagliptin DDI), subjects stayed in the clinic until 72 h post-dose.

For all Groups, blood samples for PK analysis were collected in each period prior to dosing (pre-dose) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose. For Group 3, PK blood samples were also collected at 60 and 72 h post-dose. Plasma concentrations of bexagliflozin and OHAs were determined by validated liquid chromatography tandem mass spectrometry (LC MS/MS) assays.

Urine samples for PD analysis were collected in 12 h intervals. For all Groups, urine samples were collected pre-dose (-12 to 0 h) and post-dose at 0 to 12 h, 12 to 24 h, 24 to 36 h, and 36 to 48 h. For Group 3, additional samples at 48 to 60 h and 60 to 72 h post-dose were collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2
2. Subjects who are non-smokers for at least 3 months prior to screening
3. Subjects who are willing and able to be confined to the clinical research facility as required by the protocol

Exclusion Criteria:

1. Subjects with a clinically significant history of allergy to drugs or latex.
2. Subjects with a history of alcohol or drug dependence in the past 12 months.
3. Subjects who have donated a significant amount of blood in the past 2 months
4. Female subjects who are pregnant or breastfeeding
5. Subjects who are not willing to use an adequate form of birth control during the study and for 30 days after discharge from clinic
6. Subjects who have taken an investigational drug in the past 30 days or 7 half-lives of the investigational drug, whichever is longer
7. Subjects who had previously received anti-diabetic medication, including metformin, sitagliptin, glimepiride or drugs of the same class (i.e. biguanides, DPP-4 inhibitors or sulfonylureas), or SGLT2 inhibitors, in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Chair — Massachusetts General Hospital
Locations (1):
- Clinical Research Site, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Bexagliflozin + Metformin: Bexagliflozin tablets 20 mg alone, Metformin tablets 1000 mg alone, or Bexagliflozin 20 mg + Metformin 1000 mg
- Group 2: Bexagliflozin + Glimepiride: Bexagliflozin tablets 20 mg alone, Glimepiride tablets 2 mg alone, or Bexagliflozin 20 mg + Glimepiride 2 mg
- Group 3: Bexagliflozin + Sitagliptin: Bexagliflozin tablets 20 mg alone, Sitagliptin 100 mg alone, or Bexagliflozin 20 mg + Sitagliptin 100 mg
Period: Overall Study
Arm/Group | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin + Sitagliptin
Started | 18 | 18 | 18
Completed | 18 | 18 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin + Sitagliptin | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (15.69) | 37.6 (8.25) | 43.6 (14.52) | 41.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 9 | 20
  Male | 12 | 13 | 9 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 18 | 17 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 10 | 20
  White | 13 | 12 | 8 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 79.0 (11.75) | 77.9 (12.37) | 79.0 (13.21) | 78.6 (12.23)
Height [Mean (Standard Deviation); unit: cm] | 173.3 (9.16) | 172.3 (6.45) | 170.5 (8.37) | 172.0 (8.01)

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 5 mL were be collected from a peripheral vein in each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose for Group 1 and 2. Pharmacokinetic (PK) blood samples were collected at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose for Group 3. Plasma was obtained from centrifugation, frozen and analyzed. Cmax was obtained directly from experimental observations.
Time Frame: Up to 72 hours
Population: The study was designed to evaluate the potential bexagliflozin drug interactions. Study participants were dosed with bexagliflozin alone, other drug alone or both drugs sequentially. The pharmacokinetic parameters were calculated based on the specific analyte using samples collected after dosing of the drug. Therefore, not all samples were analyzed for all outcome measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 1: Metformin Alone: Metformin: Metformin tablets, 1000 mg
- Group 1: Bexagliflozin + Metformin: Bexagliflozin: Bexagliflozin tablets, 20 mg
  Metformin: Metformin tablets, 1000 mg
- Group 2: Glimepiride Alone: Glimepiride: Glimepiride tablets, 2 mg
- Group 2: Bexagliflozin + Glimepiride: Bexagliflozin: Bexagliflozin tablets, 20 mg
  Glimepiride: Glimepiride tablets, 2 mg
- Group 3: Sitagliptin Alone: Sitagliptin: Sitagliptin tablets, 100 mg
- Group 3: Bexagliflozin + Sitagliptin: Bexagliflozin: Bexagliflozin tablets, 20 mg
  Sitagliptin: Sitagliptin tablets, 100 mg
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 18 | 18 | 18 | 18 | 18
ng/mL
  Bexagliflozin PK parameters: number analyzed (Participants) | 18 | 0 | 18 | 17 | 0 | 18 | 18 | 0 | 18
  Bexagliflozin PK parameters | 124.6 (43.7) |  | 135.5 (40.0) | 158.6 (53.9) |  | 143.7 (37.9) | 117.1 (34.6) |  | 148.3 (22.1)
  Metformin PK parameters: number analyzed (Participants) | 0 | 18 | 18 | 0 | 0 | 0 | 0 | 0 | 0
  Metformin PK parameters |  | 2067.6 (27.2) | 1965.2 (33.6) |  |  |  |  |  |
  Glimepiride PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0
  Glimepiride PK parameters |  |  |  |  | 59.9 (32.2) | 67.1 (29.5) |  |  |
  Sitagliptin PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
  Sitagliptin PK parameters |  |  |  |  |  |  |  | 356.6 (22.3) | 351.2 (32.9)
Statistical Analysis 1: Comparison: Group 1: Bexagliflozin Alone vs Group 1: Bexagliflozin + Metformin; Geometric Least Square (LS) Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 108.73, 95% CI 2-sided [94.35 to 125.30] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 2: Comparison: Group 1: Metformin Alone vs Group 1: Bexagliflozin + Metformin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 95.05, 90% CI 2-sided [84.73 to 106.63] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 3: Comparison: Group 2: Bexagliflozin Alone vs Group 2: Bexagliflozin + Glimepiride; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 89.44, 90% CI 2-sided [70.39 to 113.65] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 4: Comparison: Group 2: Glimepiride Alone vs Group 2: Bexagliflozin + Glimepiride; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 111.95, 90% CI 2-sided [97.02 to 129.19] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 5: Comparison: Group 3: Bexagliflozin Alone vs Group 3: Bexagliflozin + Sitagliptin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 126.68, 90% CI 2-sided [112.08 to 143.17] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 6: Comparison: Group 3: Sitagliptin Alone vs Group 3: Bexagliflozin + Sitagliptin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 98.48, 90% CI 2-sided [84.90 to 114.23] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect

2. Primary Outcome: Tmax (Time of Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 5 mL were collected from a peripheral vein in each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose for Group 1 and 2. PK blood samples were collected at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose for Group 3. Plasma was obtained from centrifugation, frozen and analyzed. Tmax was obtained directly from experimental observations.
Time Frame: Up to 72 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 18 | 18 | 18 | 18 | 18
hours
  Bexagliflozin PK parameters: number analyzed (Participants) | 18 | 0 | 18 | 17 | 0 | 18 | 18 | 0 | 18
  Bexagliflozin PK parameters | 4.0 [1 to 5] |  | 3.0 [1 to 5] | 8.0 [5 to 10] |  | 6.0 [5 to 10] | 3.0 [2 to 5] |  | 4.0 [2 to 5]
  Metformin PK parameters: number analyzed (Participants) | 0 | 18 | 18 | 0 | 18 | 0 | 0 | 0 | 0
  Metformin PK parameters |  | 2.5 [1 to 3] | 2.0 [1 to 5] |  | 0 [0 to 0] |  |  |  |
  Glimepiride PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0
  Glimepiride PK parameters |  |  |  |  | 5.5 [1 to 10] | 7.0 [1 to 10] |  |  |
  Sitagliptin PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
  Sitagliptin PK parameters |  |  |  |  |  |  |  | 2.5 [1 to 5] | 2.5 [1 to 6]

3. Primary Outcome: T1/2 (Apparent Terminal Elimination Half-life)
Description: Whole venous blood samples of 5 mL were collected from a peripheral vein in each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose for Group 1 and 2. PK blood samples were collected at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose for Group 3. Plasma was obtained from centrifugation, frozen and analyzed. T1/2 was obtained directly from experimental observations.
Time Frame: Up to 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Group 2: Glimepiride Alone: Glimepiride: Glimepiride tablets, 4 mg
- Group 2: Bexagliflozin + Glimepiride: Bexagliflozin: Bexagliflozin tablets, 20 mg
  Glimepiride: Glimepiride tablets, 4 mg
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 18 | 18 | 17 | 18 | 18
hours
  Bexagliflozin PK parameters: number analyzed (Participants) | 18 | 0 | 18 | 17 | 0 | 18 | 17 | 0 | 18
  Bexagliflozin PK parameters | 10.3 (30.4) |  | 7.8 (48.6) | 8.0 (33.3) |  | 7.8 (34.4) | 12.6 (48) |  | 13.3 (38.2)
  Metformin PK parameters: number analyzed (Participants) | 0 | 18 | 18 | 0 | 0 | 0 | 0 | 0 | 0
  Metformin PK parameters |  | 9.0 (31.8) | 10.2 (32.5) |  |  |  |  |  |
  Glimepiride PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0
  Glimepiride PK parameters |  |  |  |  | 7.8 (46.8) | 6.6 (57.8) |  |  |
  Sitagliptin PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
  Sitagliptin PK parameters |  |  |  |  |  |  |  | 14.3 (22.3) | 14.8 (24.5)

4. Primary Outcome: AUC0-inf (Area Under the Plasma Concentration-time Curve From Time 0 to Infinity)
Description: Whole venous blood samples of 5 mL were collected from a peripheral vein in each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h post-dose for Group 1 and 2. PK blood samples were collected at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60 and 72 h post-dose for Group 3. Plasma was obtained from centrifugation, frozen and analyzed. AUC0-inf was estimated for each subject.
Time Frame: Up to 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 18 | 18 | 18 | 18 | 18
h*ng/mL
  Bexagliflozin PK parameters: number analyzed (Participants) | 18 | 0 | 18 | 17 | 0 | 18 | 18 | 0 | 18
  Bexagliflozin PK parameters | 1154.4 (35.1) |  | 1008.6 (40.2) | 1204.9 (48.6) |  | 1162.2 (47.8) | 1011.8 (21.5) |  | 1158.1 (21.9)
  Metformin PK parameters: number analyzed (Participants) | 0 | 18 | 18 | 0 | 0 | 0 | 0 | 0 | 0
  Metformin PK parameters |  | 13351.9 (22.5) | 13784.6 (26.0) |  |  |  |  |  |
  Glimepiride PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0
  Glimepiride PK parameters |  |  |  |  | 496.1 (53.3) | 633.0 (38.5) |  |  |
  Sitagliptin PK parameters: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
  Sitagliptin PK parameters |  |  |  |  |  |  |  | 3579.6 (14.7) | 3692.8 (16.9)
Statistical Analysis 1: Comparison: Group 1: Bexagliflozin Alone vs Group 1: Bexagliflozin + Metformin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 87.36, 90% CI 2-sided [80.02 to 95.38] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 2: Comparison: Group 1: Metformin Alone vs Group 1: Bexagliflozin + Metformin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 103.24, 90% CI 2-sided [94.59 to 112.68] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 3: Comparison: Group 2: Bexagliflozin Alone vs Group 2: Bexagliflozin + Glimepiride; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Ratio of Geometric LSM = 94.46, 90% CI 2-sided [80.34 to 111.06] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 4: Comparison: Group 2: Glimepiride Alone vs Group 2: Bexagliflozin + Glimepiride; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; [Ratio of Geometric LSM] = 127.19, 90% CI 2-sided [110.33 to 146.62] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 5: Comparison: Group 3: Bexagliflozin Alone vs Group 3: Bexagliflozin + Sitagliptin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; [Ratio of Geometric LSM] = 113.09, 90% CI 2-sided [107.61 to 118.86] — Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect
Statistical Analysis 6: Comparison: Group 3: Sitagliptin Alone vs Group 3: Bexagliflozin + Sitagliptin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; [Ratio of Geometric LSM] = 103.16, 90% CI 2-sided [99.30 to 107.17]; Confidence interval from ANOVA with treatment, period, and sequence as fixed effects, and subject as a random effect

5. Secondary Outcome: Urinary Glucose Excretion up to 0-72 hr
Description: Pre-dose urine samples were collected from -12 to 0 h for baseline measurement. Subjects was instructed to empty their bladder prior to dosing. Post-dose urine was collected in 4 batches for Groups 1 and 2 at 0 to 12 h, 12 to 24 h, 24 o 36 h, and 36 to 48 h collections. Post-dose urine was collected in batches for Group 3 at 0 to 12 h, 12 to 24 h, 24 to 36 h, 36 to 48 h, 48 to 60 h and 60 to 72 h.
Time Frame: up to 0-72 hr
Population: Only subjects with data in the specific category is analyzed
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
Number analyzed (Participants) | 18 | 18 | 18 | 17 | 17 | 18 | 18 | 18 | 18
g
  0 - 12 hours: number analyzed (Participants) | 18 | 16 | 18 | 17 | 16 | 18 | 18 | 12 | 18
  0 - 12 hours | 31.57 (8.06) | 0.02 (0.01) | 26.26 (8.86) | 36.99 (14.24) | 1.26 (4.37) | 31.02 (11.19) | 29.01 (6.84) | 0.03 (0.01) | 23.94 (7.17)
  12 - 24 hours | 17.32 (11.81) | 0.04 (0.03) | 22.57 (8.29) | 26.85 (9.51) | 0.04 (0.05) | 22.59 (11.15) | 24.38 (7.92) | 0.04 (0.05) | 22.85 (9.59)
  24 - 36 hours: number analyzed (Participants) | 18 | 16 | 18 | 17 | 17 | 18 | 18 | 15 | 18
  24 - 36 hours | 23.94 (9.16) | 0.04 (0.04) | 19.50 (8.94) | 29.79 (10.24) | 0.20 (0.42) | 28.46 (11.37) | 22.31 (8.97) | 0.17 (0.56) | 24.15 (9.27)
  36 - 48 hours: number analyzed (Participants) | 18 | 18 | 18 | 17 | 17 | 18 | 18 | 17 | 18
  36 - 48 hours | 8.91 (4.97) | 0.02 (0.01) | 5.53 (4.17) | 11.03 (7.84) | 0.03 (0.01) | 9.34 (7.55) | 9.83 (6.67) | 0.03 (0.01) | 10.17 (5.23)
  48 - 60 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 15 | 18
  48 - 60 hours |  |  |  |  |  |  | 11.32 (8.09) | 0.05 (0.07) | 11.50 (7.52)
  60 - 72 hours: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 17 | 18
  60 - 72 hours |  |  |  |  |  |  | 2.67 (3.55) | 0.02 (0.01) | 2.70 (2.91)

ADVERSE EVENTS:
Time Frame: Adverse event collection began on the first clinical admission day (Day 0) and continued through D17. The subjects were actively monitored for serious adverse events for at least 14 days after discharge from the study.
Arm/Group | Group 1: Bexagliflozin Alone | Group 1: Metformin Alone | Group 1: Bexagliflozin + Metformin | Group 2: Bexagliflozin Alone | Group 2: Glimepiride Alone | Group 2: Bexagliflozin + Glimepiride | Group 3: Bexagliflozin Alone | Group 3: Sitagliptin Alone | Group 3: Bexagliflozin + Sitagliptin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/18 | 11/18 | 13/18 | 6/18 | 2/18 | 4/18 | 3/18 | 1/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Bexagliflozin Alone (N=18) | Group 1: Metformin Alone (N=18) | Group 1: Bexagliflozin + Metformin (N=18) | Group 2: Bexagliflozin Alone (N=18) | Group 2: Glimepiride Alone (N=18) | Group 2: Bexagliflozin + Glimepiride (N=18) | Group 3: Bexagliflozin Alone (N=18) | Group 3: Sitagliptin Alone (N=18) | Group 3: Bexagliflozin + Sitagliptin (N=18)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 9 (9) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Puncture site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT02956044/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT02956044/SAP_001.pdf